CLINICAL TRIAL: NCT03268174
Title: A Placebo-Controlled, Double-Blind, Bilateral Cosmetic Study With an Open Label Extension to Evaluate the Performance of a Cosmetic Product Designed to Improve the Appearance of Skin Afflicted With Mild to Moderate Atopic Dermatitis.
Brief Title: Cosmetic Study to Improve the Appearance of Skin Afflicted With Mild to Moderate Atopic Dermatitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AOB-2016-AD
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Intervention Model Description: This is a bilateral study. Each subject will apply appropriately labeled test product to the left and right arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: AO+ Mist (or placebo) are supplied in white 100mL metered spray bottles. Test products are blinded and labeled for application to the LEFT or RIGHT side of the body
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AO+Mist (Active Comparator): AO+Mist
  Interventions: Other: AO+Mist
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: AO+Mist — Subjects receive 2 bottles of product at the Baseline visit for left and right side application. One bottle will contain Placebo only, the other bottle will contain "AO+Mist".
  Label on each bottle will indicate the arm the product is to be applied to. Subjects will be instructed in the use of the spray bottle and asked to self-administer the Test Product as follows:
  * LEFT arm where skin is affected: 4 pumps of Spray which is labeled accordingly must be applied twice-a-day to the area on the arm affected by AD- once in the morning and once in the evening for 30 days.
  * RIGHT arm where skin is affected: 4pumps of Spray which is labeled accordingly must be applied twice-a-day to the area on the arm affected by AD- once in the morning and once in the evening for 30 days.
  Arms: AO+Mist
Other: Placebo — Subjects receive 2 bottles of product at the Baseline visit for left and right side application. One bottle will contain Placebo only, the other bottle will contain "AO+Mist".
  Label on each bottle will indicate the arm the product is to be applied to. Subjects will be instructed in the use of the spray bottle and asked to self-administer the Test Product as follows:
  * LEFT arm where skin is affected: 4 pumps of Spray which is labeled accordingly must be applied twice-a-day to the area on the arm affected by AD- once in the morning and once in the evening for 30 days.
  * RIGHT arm where skin is affected: 4pumps of Spray which is labeled accordingly must be applied twice-a-day to the area on the arm affected by AD- once in the morning and once in the evening for 30 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to observe the performance of a cosmetic product, AO+Mist, on the appearance of arm skin in subjects with atopic dermatitis

DETAILED DESCRIPTION:
This is a single center, double-blind, bilateral, placebo-controlled study in subjects with Atopic Dermatitis affecting both sides of the body. Up to 20 subjects will be enrolled to participate.

Subjects will undergo a 2 week washout period prior to the Baseline procedure. Follwoing the Baseline visit assessments, subjects will be asked to apply "AO+ Mist" or placebo to the affected area of the arm twice a day (morning and night) for 30 days.

After the 30 day initial study period, subjects will automatically be rolled over to participate in the extension of the trial for another 30 days using only AO+Mist on the body parts affected by Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18
2. In good general health as determined by a thorough medical history i. Visible flexural dermatitis ii. Personal history of flexural dermatitis iii. Personal history of dry skin in the past 12 months
3. Subjects should have similar presentation and severity of AD on both arms
4. Ability to comprehend and comply with study procedures
5. Agree to commit to participate in the current protocol
6. Provide written informed consent prior to any study procedure being performed (all subjects should be able to understand the informed consent form and any other documents that subjects are required to read)

Exclusion Criteria:

1. Female subjects who are pregnant or lactating or who are trying to conceive
2. Any clinically relevant abnormality identified on the screening history or any other medical condition or circumstance making the volunteer unsuitable for participation in the study
3. Any skin condition which in the investigator's opinion may interfere with the evaluation of Atopic Dermatitis
4. Severe cases of AD that present with pustules and weeping and those cases that require urgent medical attention
5. Treatment with any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the beginning of the screening period (this includes investigational formulations of marketed products, inhaled and topical drugs)
6. Hypersensitivity to AO+Mist or its components
7. Seropositive for human immunodeficiency virus (HIV) by medical history review at screening
8. Positive for Hepatitis B virus surface antigen (HBsAg) or positive Hepatitis C virus antibody (HCV Ab) by medical history review at screening
9. Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected test product non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as assessed by physical exam and appearance | Baseline-Day 30

SECONDARY OUTCOMES:
Difference in Atopic Dermatitis EASI score | Baseline-Day 30
Difference in Skindex16 Quality of Life survey | Baseline-Day 30
Difference in Skindex 16 Quality of Life Survey during Extension Period | Day 30-60
Difference in EASI score during Extension Period | Day 30-60

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Dermatology Associates of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No